CLINICAL TRIAL: NCT02904850
Title: Validation of a Kinetic Model of Erlotinib
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5615; 2013-A01122-43
Record Dates: First submitted 2014-04-03; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Lung Cancer
Keywords: Non-small cell lung cancer; locally advanced or metastatic; erlotinib monotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- group of patients: Plasma dosage of erlotinib and OSI-420
  Interventions: Biological: group of patients

INTERVENTIONS:
Biological: group of patients — Plasma dosage of erlotinib and OSI-420 is made from the blood usually taken Further information are collected in the medical record of the patient during the CT scan reassessment after collection.

SUMMARY:
Several arguments are in favor of a therapeutic monitoring for the erlotinib, therefore, a pharmacokinetic (PK) has been prepared using data from the literature. This model must be validated at concentrations achieved in practice. This is a preliminary study before the implementation of a randomized trial confirming the therapeutic monitoring of erlotinib through this model.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving treatment with erlotinib monotherapy for locally advanced or metastatic NSCLC either first line in patients with an activating mutation of the receptor EGF-R or patients with stable disease after 4 cycles of standard first-line chemotherapy with platinum or after failure of at least one prior chemotherapy regimen
* Age> 18 years
* Subject has signed an informed consent
* Treatment initiated for at least 7 days or dosage changed for at least 7 days

Exclusion Criteria:

* Contraindication to the use of drug
* Subject to exclusion period (as determined by a previous study or in progress)
* Inability to give informed information (subject in emergency situations, difficulties in understanding the subject, ...)
* Subject under judicial protection
* Subject under tutorship or curatorship
* Pregnancy (and woman of childbearing age without contraception)
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated in the care departement of the hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Difference between plasma concentrations of erlotinib concentrations observed and predictive model | 1 year

SECONDARY OUTCOMES:
Correlation of Blood levels outsized with severe side effects or compromising the vital prognosis (treatment response, adherence (assessed by the test Morisky Green) | 1 year
  Evaluation of interest to assay the active metabolite OSI-420 Observation between incidence of clinical problems (ineffectiveness, toxicity, adherence) and blood concentrations of erlotinib outsized.
  Evaluation of the potential clinical benefit to provide a dosage of erlotinib

CONTACTS AND LOCATIONS:
Overall Officials: Anne Elisabeth QUOIX, Principal Investigator — Service Pneumologie Hôpitaux Universitaires Strasbourg 67 091 STRASBOURG cedex
Locations (1):
- Service de Pneumologie Nouvel Hôpital Civil, Strasbourg, Alsace, France